CLINICAL TRIAL: NCT04425668
Title: Effect of Academic Detailing to Reduce Opioid Prescribing in Dentistry: a Randomized Quality Improvement Effort
Brief Title: Effect of Academic Detailing to Reduce Opioid Prescribing in Dentistry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Michigan Department of Health and Human Services (Other)
Responsible Party: Principal Investigator, Chad Brummett, Professor of Anesthesiology Research, Senior Associate Chair for Research, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HUM00175142
Record Dates: First submitted 2020-06-03; First posted 2020-06-11 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Opioid Prescribing; Pain Management
Keywords: Dentist
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Single blinded- dentists to be blinded; Analyses will be done by blinded analyst
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator)
  Interventions: Other: Continuing educational
- Academic detailing intervention (Experimental)
  Interventions: Behavioral: Academic detailing (AD)

INTERVENTIONS:
Behavioral: Academic detailing (AD) — In addition to continuing educational (CE) videos this group will receive up to two personalized, one-on-one, education sessions from an academic detailer. The sessions will last between 15-30 minutes. Each AD visit will consist of: an introduction, a brief needs assessment, key educational messages, a discussion of challenges the provider faces, and giving the provider leave-behind educational materials. The AD visit key educational messages are specific recommendations for opioid-prescribing practice change. When appropriate the detailer will suggest a phone call with Dr. Romesh Nalliah to discuss specific dentistry questions. There may also be a second AD visit if agreed upon by the dentist.
  Arms: Academic detailing intervention
Other: Continuing educational — Dentists enrolled in the CE program will serve as the control group. They will have access to the 3 hours of CE content online similar to the AD group; however, they will not receive academic detailing or the opportunity to connect via phone with Dr. Nalliah.
  In this group, if the dentists have content-specific questions after participating in the CE program, they may contact MichiganOPENdental@umich.edu for responses appropriately directed to Dr. Nalliah.
  Arms: Control Group

SUMMARY:
The purpose of this project is to improve quality of care for dental patients in the state of Michigan. This will be achieved through educating dentists about best practices for opioid prescribing and includes three continuing education (CE) credits and one (or two) academic detailing (AD) visits. The cohort of 90 dentists who are enrolled to the CE will be randomized into two groups upon enrollment. One of these groups, half of the cohort, will receive the academic detailing. A report will be written highlighting key findings from this project and best practices for treating patients after dental care.The quality of care for dental patients will be improved by sharing this information with both participating and non-participating dental providers statewide through reports, manuscripts, and presentations. These data will inform best practice with the potential for future academic detailing and educational interventions for dentists and oral surgeons.

ELIGIBILITY:
Inclusion Criteria:

* Dentists in the state of Michigan with an active drug enforcement agency (DEA) license.

Exclusion Criteria:

* All oral Surgeons in Michigan. Michigan dentists who have a significant (>5%) population living outside of Michigan (self-reported), as the prescription drug monitoring program (PDMP) data we will obtain from Michigan Automated Prescription Service (MAPS) will only cover those prescriptions filled in the state of Michigan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2021-05-29 (Actual); Study Completion 2021-05-29 (Actual)

PRIMARY OUTCOMES:
Change in the amount of opioid prescribed measured in the total oral morphine equivalents | baseline, up to 3 months
  Opioid data from the Michigan Automated Prescription Service (MAPS), state prescription drug monitoring program (PDMP) will be used. These periods yield 63 working weekdays in each period.

SECONDARY OUTCOMES:
Change in the number of opioid prescriptions | baseline, up to 3 months
  Number of opioid prescription details through PDMP data pulled from MAPS.

CONTACTS AND LOCATIONS:
Overall Officials: Chad Brummett, M.D., Principal Investigator — University of Michigan
Locations (1):
- Chad Brummett, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No